CLINICAL TRIAL: NCT02584140
Title: Multimodal Interventions to Improve Adherence to Oral Tenofovir/Emtricitabine as Pre-Exposure Prophylaxis in Women in Southern California
Brief Title: Pre-exposure Prophylaxis (PrEP) Adherence Enhancement Guided by iTAB and Drug Levels for Women
Acronym: AEGiS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, San Diego (Other); California HIV/AIDS Research Program (Other); Los Angeles County Department of Public Health (Other Government); AIDS Project Los Angeles (Other)
Responsible Party: Principal Investigator, Dr. Raphael Landovitz, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-001583
Record Dates: First submitted 2015-10-15; First posted 2015-10-22 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: HIV Prevention
Keywords: PrEP; Pre-exposure Prophylaxis; HIV Prevention

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive daily oral emtricitabine/tenofovir disoproxil fumarate, adherence counseling, and daily text message reminders.
Oversight: Data Monitoring Committee: No

ARMS (1):
- AEGIS (Other): All participants will be assigned to this arm of the study.
  Interventions: Behavioral: Text Messaging; Behavioral: Adherence Counseling; Drug: Daily Oral PrEP

INTERVENTIONS:
Behavioral: Text Messaging — All participants assigned to the iTAB intervention will receive daily dosing reminders that will be sent for the first 6 weeks and then continue with reminders for the duration of the study.
  Other Names: iTAB
Behavioral: Adherence Counseling — All participants assigned to the counseling intervention will receive sexual health and medication adherence counseling at each study visit. Participants with suboptimal adherence (TFV-DP levels of <1050 fmol/punch (representing fewer than mean 6-7 daily doses per week)) will trigger a targeted iNSC session. Participants with two TFV-DP levels of <1050 fmol/punch will trigger PrEP Steps, a higher intensity adherence counseling intervention consisting of four 50-minute counseling sessions and 2 booster counseling sessions.
  Other Names: Integrate Next Step Counseling (iNSC); Targeted iNSC; PrEP Steps
Drug: Daily Oral PrEP — All participants will be offered daily oral emtricitabine/tenofovir disoproxil fumarate for Pre-exposure Prophylaxis.
  Other Names: PrEP

SUMMARY:
The purpose of this study is to test a program that uses drug level monitoring, text messaging ("iTAB") and personalized counseling with HIV prevention services, including PrEP (medicine that can help prevent HIV infection when taken daily).

DETAILED DESCRIPTION:
This is an open-label single-arm longitudinal clinical trial to estimate medication adherence and retention in a PrEP HIV prevention program that implements a combination intervention strategy that uses text-messages (iTAB) and a staged adherence counseling support strategy titrated from real-time drug levels in women at-risk for HIV acquisition.

A total of 135 participants will receive the combined intervention of text messaging adherence reminders and adherence support. The text messaging system consists of daily, personalized, automated 2-way text messages to maintain adherence and retention. Participants that have a low intracellular tenofovir diphosphate (TFV-DP) concentration will receive escalated, targeted adherence support. All participants will receive access to PrEP in accordance with standardized comprehensive methods of prescribing and clinical assessments that include safety monitoring as well as regular HIV and sexually transmitted infection (STI) screening. All participants will be followed for 48 weeks after enrollment and will receive a post study follow-up at 60 weeks. The primary endpoint will be measured at 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth and identifies as female gender
* Age 18 years or older
* Able to understand and provide consent in English or Spanish
* HIV negative by 4th generation test (Ag/Ab test) or combination of enzymeimmunoassay (EIA) and HIV RNA
* Creatinine clearance ≥ 60 ml/min (via Cockcroft-Gault formula)

At-Risk Criteria (at least one):

* Condomless sex in the last 3 months with one or more male partners of unknown HIV status known to be at substantial risk of HIV infection (IDU, bisexual, sex for goods, recently incarcerated, from a country with HIV prevalence >1%, interpersonal Partner Violence);
* STI (rectal or vaginal gonorrhea or syphilis) diagnosis during the last 6 months.
* Previous post-exposure prophylaxis (PEP) use during the last 12 months.
* Has at least one HIV-infected sexual partner for ≥4 weeks.
* Sex for exchange of money, goods or services

Exclusion Criteria:

* Pregnancy at enrollment.
* Any condition, which in the opinion of the provider, will seriously compromise the participant's ability to comply with the protocol, including adherence to PrEP medication dosing, such as active, untreated or unstable major mental illness (i.e. untreated psychotic disorder).
* Use of prohibited medications, in particular, agents known to be nephrotoxic or drugs slow in renal excretion.
* Previous participation in an HIV vaccine trial. Participants that were documented to have received only placebo are not excluded.
* Signs or symptoms suspicious for Primary HIV Infection (PHI).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Landovitz, MD, Principal Investigator — University of California, Los Angeles; Sheldon Morris, MD, Principal Investigator — UCSD
Locations (5):
- United States (5):
  - APLA Health & Wellness' Gleicher / Chen Health Center, Los Angeles, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA, Los Angeles, California
  - USC 5P21 Rand Schrader Clinic, Los Angeles, California
  - T.H.E. at Ruth Temple, Los Angeles, California
  - UCSD Antiviral Research Center, San Diego, California

REFERENCES:
- [Derived] Anderson KM, Blumenthal J, Jain S, Sun X, Amico KR, Landovitz R, Zachek CM, Morris S, Moore DJ, Stockman JK. The impact of intimate partner violence on PrEP adherence among U.S. Cisgender women at risk for HIV. BMC Public Health. 2024 May 31;24(1):1461. doi: 10.1186/s12889-024-18946-4. PMID 38822300
- [Derived] Blumenthal J, Landovitz R, Jain S, He F, Kofron R, Ellorin E, Ntim GM, Stockman JK, Corado K, Rivet Amico K, Moore DJ, Morris S. Pre-Exposure Prophylaxis Perspectives, Sociodemographic Characteristics, and HIV Risk Profiles of Cisgender Women Seeking and Initiating PrEP in a US Demonstration Project. AIDS Patient Care STDS. 2021 Dec;35(12):481-487. doi: 10.1089/apc.2021.0114. PMID 34851726

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AEGIS
Started | 136
Completed | 83
Not Completed | 53

BASELINE CHARACTERISTICS:
Arm/Group | AEGIS
Number analyzed (Participants) | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.16 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 30
  Non-Hispanic Black | 52
  Latina | 26
  Other | 28
Region of Enrollment [Number; unit: participants]
  United States | 136
Education [Count of Participants; unit: Participants]
  High school or less | 61
  Some college or more | 75
Monthly Income [Count of Participants; unit: Participants]
  $2,000 or less | 74
  More than $2,000 | 35
  No response | 27
Relationship [Count of Participants; unit: Participants]
  Divorced/Widowed/Separated | 17
  Married/Monogamous | 53
  Single/Open | 63
  No response | 3
Employment [Count of Participants; unit: Participants]
  Full/Part time/Retired | 68
  Unemployed/Unable to work | 60
  No response | 8

OUTCOME MEASURES:

1. Primary Outcome: Adherence to PrEP
Description: Adherence is measured by TFV-DP (tenofovir diphosphate) concentrations in Dried Blood Spots (DBS) suggestive of 6-7 doses per week.
Time Frame: Week 4 to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | AEGIS
Number analyzed (Participants) | 136
Participants
  Week 4: <2 doses (BLQ - 349 fmol/punch) | 22
  Week 4: 2-3 doses (350 - 699 fmol/punch) | 11
  Week 4: 4-5 doses (700 - 1049 fmol/punch) | 30
  Week 4: 6-7 doses (≥ 1050 fmol/punch) | 54
  Week 4: Missed Visit, Withdrawal, Off PrEP | 19
  Week 12: <2 doses (BLQ - 349 fmol/punch) | 21
  Week 12: 2-3 doses (350 - 699 fmol/punch) | 19
  Week 12: 4-5 doses (700 - 1049 fmol/punch) | 17
  Week 12: 6-7 doses (≥ 1050 fmol/punch) | 45
  Week 12: Missed Visit, Withdrawal, Off PrEP | 34
  Week 24: <2 doses (BLQ - 349 fmol/punch) | 15
  Week 24: 2-3 doses (350 - 699 fmol/punch) | 11
  Week 24: 4-5 doses (700 - 1049 fmol/punch) | 25
  Week 24: 6-7 doses (≥ 1050 fmol/punch) | 29
  Week 24: Missed Visit, Withdrawal, Off PrEP | 56
  Week 36: <2 doses (BLQ - 349 fmol/punch) | 16
  Week 36: 2-3 doses (350 - 699 fmol/punch) | 8
  Week 36: 4-5 doses (700 - 1049 fmol/punch) | 17
  Week 36: 6-7 doses (≥ 1050 fmol/punch) | 28
  Week 36: Missed Visit, Withdrawal, Off PrEP | 67
  Week 48: <2 doses (BLQ - 349 fmol/punch) | 16
  Week 48: 2-3 doses (350 - 699 fmol/punch) | 8
  Week 48: 4-5 doses (700 - 1049 fmol/punch) | 17
  Week 48: 6-7 doses (≥ 1050 fmol/punch) | 25
  Week 48: Missed Visit, Withdrawal, Off PrEP | 70

2. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events
Description: Describe the safety and tolerability of daily emtricitabine/tenofovir disoproxil fumarate TDF/FTC given for PrEP including discontinuation for any adverse event, serious adverse events and adverse events (grade 2 or higher).
Time Frame: Baseline to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | AEGIS
Number analyzed (Participants) | 136
Participants
  One of more grade 2+ AEs | 72
  No grade 2+ AEs reported | 64

3. Secondary Outcome: Number of HIV Infections
Description: Number of new HIV infections observed among participants with at least one follow-up visit.
Time Frame: Baseline to Week 48
Population: Participants with one or more follow-up visits were included in this analysis
Measure: Number; unit: infections
Arm/Group | AEGIS
Number analyzed (Participants) | 121
infections | 0

4. Secondary Outcome: Correlates of PrEP Adherence
Description: Self-reported adherence by daily texting through iTAB will be correlated with TFV-DP concentrations in DBS
Time Frame: Baseline to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | AEGIS
Number analyzed (Participants) | 136
Participants
  Week 4: TFV-DP <1050 fmol/punch (0-5 doses weekly) | 58
  Week 4: TFV-DP ≥1050 fmol/punch (6-7 doses weekly) | 50
  Week 4: Missing/Withdrawn/On study, off medication | 28
  Week 12: TFV-DP <1050 fmol/punch (0-5 doses weekly) | 55
  Week 12: TFV-DP ≥1050 fmol/punch (6-7 doses weekly) | 44
  Week 12: Missing/Withdrawn/On study, off medication | 37
  Week 24: TFV-DP <1050 fmol/punch (0-5 doses weekly) | 48
  Week 24: TFV-DP ≥1050 fmol/punch (6-7 doses weekly) | 28
  Week 24: Missing/Withdrawn/On study, off medication | 60
  Week 36: TFV-DP <1050 fmol/punch (0-5 doses weekly) | 39
  Week 36: TFV-DP ≥1050 fmol/punch (6-7 doses weekly) | 26
  Week 36: Missing/Withdrawn/On study, off medication | 71
  Week 48: TFV-DP <1050 fmol/punch (0-5 doses weekly) | 38
  Week 48: TFV-DP ≥1050 fmol/punch (6-7 doses weekly) | 23
  Week 48: Missing/Withdrawn/On study, off medication | 75
Statistical Analysis 1: Comparison: AEGIS; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — The P-Value for Week 4 was <0.001; The P-Value for Week 12 was 0.005; The P-Value for Week 24 was 0.029; The P-Value for Week 36 was 0.008; The P-Value for Week 48 was 0.03

ADVERSE EVENTS:
Time Frame: 48 Weeks
Arm/Group | AEGIS
All-Cause Mortality (participants affected / at risk) | 0/136
Serious Adverse Events (participants affected / at risk) | 0/136
Other Adverse Events (participants affected / at risk) | 64/136
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEGIS (N=136)
Headache (Nervous system disorders) | 4 (4)
Abdominal Discomfort (Gastrointestinal disorders) | 5 (5)
Decreased Creatinine Clearance (Investigations) | 61 (126)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT02584140/Prot_SAP_000.pdf